CLINICAL TRIAL: NCT02727322
Title: A Randomized, Double-blind, Placebo-controlled Trial of Nitrofurantoin Prophylaxis During Catheterization for Acute Postoperative Urinary Retention After Pelvic Reconstructive Surgery
Brief Title: Nitrofurantoin Prophylaxis During Catheter-managed Acute Urinary Retention After Pelvic Reconstructive Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Halina M Zyczynski, MD (Other)
Responsible Party: Sponsor-Investigator, Halina M Zyczynski, MD, Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PRO15110557
Record Dates: First submitted 2016-03-31; First posted 2016-04-04 (Estimated); Results first posted 2019-05-20 (Actual); Last update posted 2019-05-29 (Actual); Status verified 2019-05

CONDITIONS: Pelvic Organ Prolapse
MeSH Terms: conditions — Pelvic Organ Prolapse | interventions — Nitrofurantoin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nitrofurantoin (Active Comparator): Receives once daily nitrofurantoin 100mg
  Interventions: Drug: Nitrofurantoin
- Placebo (Placebo Comparator): Receives matching placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Nitrofurantoin — Patients will receive nitrofurantoin 100mg once daily or a placebo. Pills will be identical.
  Other Names: Macrobid
  Arms: Nitrofurantoin
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The specific aim of this randomized double-blind placebo-controlled trial is to determine if extended release nitrofurantoin antibiotic prophylaxis decreases the incidence of symptomatic urinary tract infection (UTI) compared with placebo for patients undergoing short term indwelling or clean intermittent self-catheterization (CISC) for acute postoperative urinary retention following pelvic organ prolapse and/or urinary incontinence surgery.

Consented patients who undergo urogenital surgery and fail their post-operative voiding trial will be randomized to either extended release nitrofurantoin 100mg or an identical appearing placebo capsule to be taken daily while performing CISC or while indwelling catheter is in place. The primary outcome will be symptomatic and culture confirmed UTI within six weeks of surgery. Secondary outcomes include adverse events associated with nitrofurantoin use, and incidence of nitrofurantoin-resistant isolates from urine culture of symptomatic women.

Primary and secondary outcomes will be evaluated with Student t test and chi squared or Fisher exact test as appropriate. Assuming a decrease in symptomatic UTIs attributable to nitrofurantoin prophylaxis from 33% to 13%, with 80% power, and a two-sided alpha of 0.05, and a 10% dropout rate, we should recruit a total of 154 patients.

DETAILED DESCRIPTION:
Urinary tract infections (UTI) occur frequently following surgery for urinary incontinence or pelvic organ prolapse (POP), with reported incidence up to 48%. This high rate is frequently attributed to intraoperative factors, such as manipulation of the genitourinary tract and instrumentation of the bladder and urethra, as well as an approximately 50% rate of short term postoperative catheterization following urogynecologic surgery. As American women have a 20% lifetime risk of surgery for POP or urinary incontinence, the absolute number of women at risk for urinary infectious morbidity associated with these procedures is quite high.

The substantial risk of UTI following POP or incontinence surgery, combined with the well-established risk associated with catheterization, leads many practitioners to prescribe oral antibiotics to women undergoing catheterization in the postoperative period. However, there is minimal Level I evidence to support or refute this practice. The Infectious Disease Society of America (IDSA) Guideline acknowledges that prophylactic antibiotics have been shown to reduce UTI rates among patients using short term postoperative catheterization in randomized trials. However, they recommend against routine antibiotic prophylaxis use due to concerns regarding anti-microbial resistance, cost, and potential for adverse effects, even among high risk groups including women undergoing urogynecologic surgery. This recommendation is based on expert opinion, given a paucity of trial data to guide clinical care.

Nitrofurantoin is a commonly used antibiotic for UTI prophylaxis during catheterization, is well-tolerated with few adverse effects, and is known to have a very low rate of associated resistance. After decades of use, it remains active against the most common UTI pathogens that have gained resistance to other antimicrobials. For example, in the 2013 Magee-Womens Hospital Adult Antibiogram, 98% of E-coli specimens were sensitive to Nitrofurantoin, which has been consistent since at least 2007. The drug has a half-life of 20 minutes and 40% is concentrated in and excreted into the urine in a therapeutically unchanged form. Thus it has minimal impact on vaginal and bowel flora. Nitrofurantoin has been shown to reduce the incidence of positive urine cultures and symptomatic UTIs in women with a suprapubic catheter after pelvic organ prolapse and/or urinary incontinence surgery. No trials have evaluated nitrofurantoin prophylaxis for women using short term indwelling catheters or CISC following urogynecologic procedures.

Given the large number of women at risk for urinary infectious morbidity associated with short term catheterization for acute urinary retention following POP and/or incontinence surgery, and the paucity of data on the impact of antibiotic prophylaxis in this setting, we propose to demonstrate the efficacy of nitrofurantoin prophylaxis through an adequately-powered, placebo-controlled trial. Secondary outcomes will include adverse events associated with nitrofurantoin use, and incidence of nitrofurantoin resistant bacterial isolates from urine culture.

Primary Aim: To determine if extended release nitrofurantoin administered daily to patients using indwelling or clean intermittent self-catheterization (CISC) after pelvic organ prolapse and/or urinary incontinence surgery will decrease the incidence of symptomatic and culture proven urinary tract infection (UTI) when compared to placebo in a randomized, double-blind trial.

Secondary Aim(s): To determine how nitrofurantoin antibiotic prophylaxis administered to patients using an indwelling catheter or CISC after pelvic organ prolapse and/or urinary incontinence surgery affects frequency of adverse events related to daily nitrofurantoin exposure, and frequency of urine cultures positive for nitrofurantoin-resistant isolates.

The Null Hypotheses: Nitrofurantoin antibiotic prophylaxis administered to patients using an indwelling catheter or CISC after pelvic organ prolapse and/or urinary incontinence surgery does not change the incidence of symptomatic and culture proven urinary tract infection (UTI) compared with placebo.

ELIGIBILITY:
Inclusion Criteria:

- Women who have undergone surgery for the correction of pelvic organ prolapse and/or urinary incontinence and failed a postoperative voiding trial

Exclusion Criteria:

* Known drug allergy to nitrofurantoin
* History of renal insufficiency
* Renal transplant
* Renal nephropathy
* Recent history of more than 3 UTIs per year
* History of nitrofurantoin-induced pulmonary injury or nitrofurantoin associated cholestatic jaundice/hepatic dysfunction
* Known immunocompromised condition (organ transplant, chemotherapy, immune suppression associated with autoimmune disease).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2016-08; Primary Completion 2018-03-27 (Actual); Study Completion 2018-05-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Erin S Lavelle, MD, Principal Investigator — University of Pittsburgh
Locations (2):
- United States (2):
  - Georgetown/MedStar Hospital Center, Washington D.C., District of Columbia
  - Magee-Womens Hospital of UPMC, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No
No plan to make participant data available

REFERENCES:
- [Derived] Lavelle ES, Alam P, Meister M, Florian-Rodriguez M, Elmer-Lyon C, Kowalski J, Carter-Brooks C, Mazloomdoost D, Zyczynski H, Lowder J, Gutman R, Sutkin G. Antibiotic Prophylaxis During Catheter-Managed Postoperative Urinary Retention After Pelvic Reconstructive Surgery: A Randomized Controlled Trial. Obstet Gynecol. 2019 Oct;134(4):727-735. doi: 10.1097/AOG.0000000000003462. PMID 31503155

RESULTS

PARTICIPANT FLOW:
Groups:
- Nitrofurantoin: Receives once daily nitrofurantoin 100mg
  Nitrofurantoin: Patients will receive nitrofurantoin 100mg once daily during catheter use.
- Placebo: Receives matching placebo
  Placebo: Patients will receive identical appearing placebo once daily during catheter use.
Period: Overall Study
Arm/Group | Nitrofurantoin | Placebo
Started | 77 | 77
Completed | 75 | 76
Not Completed | 2 | 1
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Population: Does not include 3 participants withdrawn.
Groups:
- Total: Total of all reporting groups
Arm/Group | Nitrofurantoin | Placebo | Total
Number analyzed (Participants) | 75 | 76 | 151
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.7 (11.9) | 60.5 (12.0) | 60.9 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 75 | 76 | 151
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 64 | 60 | 124
  African American | 5 | 11 | 16
  Native American | 1 | 1 | 2
  Hispanic | 5 | 4 | 9
Body Mass Index (kg/m^2) [Mean (Standard Deviation); unit: kg/m^2] | 26.8 (4.4) | 27.5 (5.3) | 27.2 (5.1)
Gravidity [Mean (Standard Deviation); unit: number of pregnancies] | 3 (2) | 3 (2) | 3 (2)
Parity [Mean (Standard Deviation); unit: pregnancies delivered after 20 weeks] | 3 (1) | 3 (1) | 3 (1)
Current Smoker [Count of Participants; unit: Participants] | 4 | 3 | 7
Menopausal Status [Count of Participants; unit: Participants]
  Premenopausal | 15 | 17 | 32
  Postmenopausal, No Hormone Replacement therapy | 56 | 57 | 113
  Postmenopausal, Oral Hormone Replacement Therapy | 4 | 2 | 6
Vaginal Estrogen Use [Count of Participants; unit: Participants] | 20 | 22 | 42
Diabetes, on medication [Count of Participants; unit: Participants] | 4 | 9 | 13
History of Urinary Tract Infection in past year [Count of Participants; unit: Participants] | 2 | 6 | 8
Preoperative POP-Q Stage [Count of Participants; unit: Participants] — POP-Q is a measure of the degree of Pelvic Organ Prolapse present. Stage 0 is essentially no prolapse or descent of pelvic organs; higher stages indicate progressively larger degrees of prolapse.
  Participants
    0 | 2 | 3 | 5
    1 | 4 | 6 | 10
    2 | 27 | 16 | 43
    3 | 38 | 37 | 75
    4 | 1 | 5 | 6
    unknown | 3 | 9 | 12
Preoperative Postvoid Residual Volume [Mean (Standard Deviation); unit: ml] | 87.4 (147.5) | 66.4 (129.4) | 72.8 (95.3)
Indication for surgery [Count of Participants; unit: Participants]
  Prolapse | 38 | 31 | 69
  Incontinence | 12 | 19 | 31
  Prolapse and Incontinence | 25 | 26 | 51

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing Urinary Tract Infection Within 6 Weeks of Surgery
Description: Frequency of symptomatic, culture-proven UTI; included participants who were empirically treated outside of protocol (symptoms but no culture) within 6 weeks of surgery.
  Positive culture was defined as at least 100,000 colony forming units (cfu)/ml of uropathic bacteria in a catheterized or midstream clean catch voided urine specimen.
Time Frame: within 6 weeks of surgery
Measure: Count of Participants; unit: Participants
Groups:
- Nitrofurantoin: Receives once daily nitrofurantoin 100mg
  Nitrofurantoin: Patients will receive nitrofurantoin 100mg once daily during catheterization.
- Placebo: Receives matching placebo
  Placebo: Patients will receive identical appearing placebo daily during catheterization.
Arm/Group | Nitrofurantoin | Placebo
Number analyzed (Participants) | 75 | 76
Participants | 13 | 13
Statistical Analysis 1: Comparison: Nitrofurantoin vs Placebo; Test type: Superiority; p = 0.97, Chi-squared; Risk Ratio (RR) = 1.1, 95% CI 2-sided [0.50 to 2.04]

2. Secondary Outcome: Number of Participants Who Experienced at Least One Adverse Event Symptom While Requiring Catheterization
Description: This is the number of participants who experienced at least one adverse symptom as reported on the diary completed daily while requiring catheterization. These adverse symptoms included: constipation, nausea/vomiting, drowsiness, headache, flatulence, abdominal pain, dizziness, diarrhea, rash/itching, dyspepsia, fever/chills, amblyopia and other.
Time Frame: within 6 weeks of surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Nitrofurantoin | Placebo
Number analyzed (Participants) | 75 | 76
Participants | 51 | 46
Statistical Analysis 1: Comparison: Nitrofurantoin vs Placebo; Test type: Superiority; p = 0.665, Chi-squared; Risk Ratio (RR) = 1.12, 95% CI 2-sided [0.885 to 1.43]

3. Secondary Outcome: Frequency of Urine Cultures Positive for Nitrofurantoin-resistant Isolates
Description: Frequency of urine cultures with one or more organisms resistant to nitrofurantoin. Positive culture was defined as at least 100,000 colony forming units (cfu)/ml of uropathic bacteria in a catheterized or midstream clean catch voided urine specimen.
Time Frame: within 6 weeks of surgery
Measure: Number; unit: nitrofurantoin resistant urine cultures
Units Other Than Participants: Positive urine cultures
Arm/Group | Nitrofurantoin | Placebo
Number analyzed (Participants) | 75 | 76
Number analyzed (Positive urine cultures) | 12 | 15
nitrofurantoin resistant urine cultures | 4 | 3
Statistical Analysis 1: Comparison: Nitrofurantoin vs Placebo; Test type: Superiority; p = 1.0, Fisher Exact; Risk Ratio (RR) = 1.32, 95% CI 2-sided [0.31 to 5.68]

ADVERSE EVENTS:
Time Frame: 6 weeks since randomization
Description: Participants completed daily diaries during catheterization in which they reported adverse effects. Study coordinators also solicited adverse events from participants at 6 weeks, and reviewed medical records for adverse events.
Arm/Group | Nitrofurantoin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/75 | 0/76
Serious Adverse Events (participants affected / at risk) | 3/75 | 2/76
Other Adverse Events (participants affected / at risk) | 18/75 | 16/76
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nitrofurantoin (N=75) | Placebo (N=76)
Transient Ischemic Attack (Vascular disorders) | 0 (0) | 1 (1)
Transfusion (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Voiding Dysfunction Requiring Surgery (Renal and urinary disorders) | 2 (2) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nitrofurantoin (N=75) | Placebo (N=76)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
Lower Extremity Symptoms (Nervous system disorders) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2)
Dysuria (Renal and urinary disorders) | 1 (1) | 2 (2)
Hematuria (Renal and urinary disorders) | 3 (3) | 1 (1)
Prolonged Urinary Retention (Renal and urinary disorders) | 1 (1) | 2 (2)
Catheter Discomfort or Obstruction (Renal and urinary disorders) | 3 (3) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Infection of Incision (Infections and infestations) | 2 (2) | 3 (3)
Vulvovaginal Yeast Infection (Infections and infestations) | 1 (1) | 0 (0)
Infected Hematoma (Infections and infestations) | 1 (1) | 0 (0)
(General disorders) | 0 (0) | 2 (2)

LIMITATIONS AND CAVEATS:
The per protocol analysis did not meet power. Not powered for secondary outcomes - antibiotic resistance and adverse symptoms.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-11-01): https://cdn.clinicaltrials.gov/large-docs/22/NCT02727322/Prot_SAP_000.pdf